CLINICAL TRIAL: NCT00582998
Title: Vacuum Assisted Closure as a Treatment for Soft Tissue Injuries Sustained as a Result of Calcaneus, Tibial Plateau and Pilon Fractures
Brief Title: Vacuum Assisted Closure as a Treatment for Soft Tissue Injuries
Acronym: VAC-ST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Principal Investigator, Steven Theiss, MD, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F010316003
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-05

CONDITIONS: Fracture of Calcaneus, Pilon or Tibial Plateau
Keywords: Vacuum Assisted Closure (VAC); Calcaneus Fracture; Pilon Fracture; Tibial Plateau Fracture; Open Reduction and Internal Fixation
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Wound Dressing (Active Comparator): Standard post-operative wound dressing
  Interventions: Procedure: Standard Wound Dressing
- Vacuum Assisted Closure Device (Active Comparator): Vacuum Assisted Closure (VAC) device
  Interventions: Device: Vacuum Assisted Closure Device

INTERVENTIONS:
Procedure: Standard Wound Dressing — Following repair of fracture of calcaneus, pilon or tibial plateau, a standard wound dressing is applied in the OR. Dressing is taken down post-op day 1 to evaluate draining, and if necessary, replaced. Dressing will be monitored for drainage every 48 hours until wound is clean, dry and intact.
  Arms: Standard Wound Dressing
Device: Vacuum Assisted Closure Device — Following repair of fracture of calcaneus, pilon or tibial plateau, a Vacuum Assisted Closure (VAC) device is applied in the OR. VAC cannister is evaluated for drainage, and if necessary, replaced. VAC sponge will be monitored for drainage every 48 hours, replaced if needed, until wound is clean, dry and intact.
  Other Names: Vacuum Assisted Closure (VAC) device
  Arms: Vacuum Assisted Closure Device

SUMMARY:
This project is designed as a prospective, randomized, comparative study evaluating the use of a negative pressure vacuum device in treating soft tissue injuries and the surgical incision following open reduction and internal fixation of calcaneus, tibial plateau, and pilon fractures.

DETAILED DESCRIPTION:
Patients who have a calcaneus fracture requiring open reduction and internal fixation through a lateral approach and who give informed consent to enter the study will be randomized into two groups. Randomization will be stratified for each of the three fracture types. Group A will be patients treated with daily dressing changes and wound evaluations beginning on post operative day 1. Group B patients will have a VAC device placed in the operating room, with the first post-operative wound evaluation taking place 48 hours post-op. If at the first post-operative evaluation there is marked drainage, the VAC device will be replaced with re-evaluation approximately 48 hours later.

The outcome variables consist of the number of days and amount of wound drainage, incidence of wound breakdown, incidence of flap coverage, incidence of infection, return to the operating room for repeat irrigation and debridement , the need for repeat wound closure, and any other intraoperative and postoperative complications recorded in medical record and on the study data collection form.

Patients who have a tibial plateau fracture requiring open reduction and internal fixation and who give informed consent to enter the study will be randomized into two groups. Group A will be patients treated with daily dressing changes and wound evaluations beginning on post operative day 2. Group B patients will have a VAC device placed in the operating room, with the first post-operative wound evaluation taking place 48 hours post-op. If at the first post-operative evaluation there is marked drainage the VAC device will be replaced with re-evaluation approximately 48 hours later. Patients with open tibial plateau fractures will be included in both groups A and B but will be sub-stratified within each group.

The outcome variables consist of the number of days and amount of wound drainage, incidence of wound breakdown, incidence of flap coverage, incidence of infection, return to the operating room for repeat irrigation and debridement , the need for repeat wound closure, and any other intraoperative and postoperative complications recorded in medical record and on the study data collection form.

Patients who have a pilon fracture requiring open reduction and internal fixation and who give informed consent to enter the study will be randomized into two groups. Group A will be patients treated with daily dressing changes and wound evaluations beginning on post operative day 2. Group B patients will have a VAC device placed in the operating room, with the first post-operative wound evaluation taking place 48 hours post-op. If at the first post-operative evaluation there is marked drainage the VAC device will be replaced with re-evaluation approximately 48 hours later. Patients with open pilon fractures will be included in both groups A and B but will be sub-stratified within each group.

The outcome variables consist of the number of days and amount of wound drainage, incidence of wound dehiscence, incidence of flap coverage, incidence of infection, return to the operating room for repeat irrigation and debridement, the need for repeat wound closure, and any other intraoperative and postoperative complications recorded in medical record and on the study data collection form. All patients will have their total lymphocyte counts and their albumin levels recorded on admission to document their nutritional status and ability to heal wounds.

Clinical photographs of the wounds will be taken with a digital camera at the time of admission to the study, and during each subsequent trip to the operating room. We will also record the injury severity score for all multiple trauma patients recorded at the time of injury in the medical record and on the study data collection form. The soft tissue score, according to the Tscherne classification for closed injuries or according to the Gustillo and Anderson classification for open injuries will also be recorded, for all multiple trauma patients, at the time of injury in the medical record and on the study data collection form. The effects will be measured by clinical examination and will be augmented with culture data for any wounds that require surgical intervention. All patients in the Intensive Care Units will have daily weights, fluid balances, and nutritional intake recorded per ICU protocol. Resuscitation data, including total fluids, blood products, and base deficit will be recorded. Fluids and blood utilization in the OR will also be documented.

The following methods and tools will be used to document study data points: intraoperative and postoperative adverse device effects recorded in the medical record and on the study data collection form, daily wound drainage as documented on rounds and in the medical record, admission total lymphocyte count and serum albumin levels, clinical evidence of infection and supplementary lab data. All of this data will be documented on the study data collection form. Patients will be followed clinically for 12 months, documenting any complications that occur with the wound (infection, dehiscence, etc…) on the study data collection form. The soft tissue score according to Tscherne classification for closed injuries, and the Gustillo and Anderson score for open injuries, will be recorded in the medical record and on the study data collection form.

Data will be collected and entered into EXCEL spreadsheets with double keying for quality control purposes and managed by the Department of Orthopaedic Surgery at the University of Alabama at Birmingham (UAB). After data entry is complete, the file(s) will be copied to diskette and delivered to the UAB Biostatistics statistician for analysis and report generation. The analysis will involve simple descriptive statistics (means, standard deviations, proportions) to assure balance of the treatment groups with respect to relevant variables. T-test will be used to compare the mean times to wound closure as well as the need for surgical debridement of the wound. Analysis of covariance will be performed if there are variables that require adjustment. Growth curve analysis (survival models) and Cox regression procedures will be used to compare the rates of wound closure between the two groups. Assumption of proportional hazards in the model will be verified before attempting Cox regression procedures. P-values will be computed using a Mann-Whitney U test for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a closed calcaneus, tibial plateau or pilon fracture requiring open reduction and internal fixation.
* Adult patients (19 years and older)

Exclusion Criteria:

* No clinical evidence of infection
* Patients unable or unwilling to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2001-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Theiss, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Background] Tarkin IS, Clare MP, Marcantonio A, Pape HC. An update on the management of high-energy pilon fractures. Injury. 2008 Feb;39(2):142-54. doi: 10.1016/j.injury.2007.07.024. Epub 2007 Dec 3. PMID 18054017
- [Background] Thompson JT, Marks MW. Negative pressure wound therapy. Clin Plast Surg. 2007 Oct;34(4):673-84. doi: 10.1016/j.cps.2007.07.005. PMID 17967622

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some of the participants had multiple fractures (there were a total of 263 fractures and 249 participants). The numbers reflected in the Participant Flow, Baseline Characteristics, and Adverse Events sections reflect participants and not fractures.
Units Other Than Participants: Fractures
Groups:
- Vacuum Assisted Closure Device: Vacuum Assisted Closure (VAC) device
  VAC: Following repair of fracture of calcaneus, pilon or tibial plateau, a Vacuum Assisted Closure (VAC) device is applied in the OR. VAC cannister is evaluated for drainage, and if necessary, replaced. VAC sponge will be monitored for drainage every 48 hours, replaced if needed, until wound is clean, dry and intact.
Period: Overall Study
Arm/Group | Standard Wound Dressing | Vacuum Assisted Closure Device
Started | 119; 122 Fractures | 130; 141 Fractures
Completed | 119; 122 Fractures | 130; 141 Fractures
Not Completed | 0; 0 Fractures | 0; 0 Fractures

BASELINE CHARACTERISTICS:
Population: The numbers reflected in the Participant Flow, Baseline Characteristics, and Adverse Events sections reflect participants and not fractures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Wound Dressing | Vacuum Assisted Closure Device | Total
Number analyzed (Participants) | 119 | 130 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 117 | 224
  >=65 years | 12 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 87
  Male | 77 | 85 | 162
Region of Enrollment [Number; unit: participants]
  United States | 119 | 130 | 249

OUTCOME MEASURES:

1. Primary Outcome: Healing of Orthopaedic Trauma Extremity Wound Fractures (Calcaneus, Pilon and Tibial Plateau)
Description: Healing of Orthopaedic Trauma Extremity Wounds: Calcaneus, Pilon and Tibial Plateau Fractures with standard dressing versus negative pressure wound therapy
Time Frame: The time from injury from surgical stabilization (14 days)
Population: as for baseline characteristics
Measure: Count of Units; unit: Fractures
Units Other Than Participants: Fractures
Arm/Group | Standard Wound Dressing | Vacuum Assisted Closure Device
Number analyzed (Participants) | 119 | 130
Number analyzed (Fractures) | 122 | 141
Fractures | 99 | 127

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Wound Dressing | Vacuum Assisted Closure Device
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/130
Other Adverse Events (participants affected / at risk) | 23/119 | 14/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Wound Dressing (N=119) | Vacuum Assisted Closure Device (N=130)
Adverse Event (Infections and infestations) | 23 (23) | 14 (14) — Post operative infection noted
Wound Dehiscence (Surgical and medical procedures) | 20 (20) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No